CLINICAL TRIAL: NCT06684158
Title: Mecapegfilgrastim Combined With Adebrelimab and Chemotherapy as Neoadjuvant Therapy in Resectable GC/GEJC: A Prospective, Randomized, Multicenter, Phase 2 Study.
Brief Title: Mecapegfilgrastim Combined With Adebrelimab and Chemotherapy as Neoadjuvant Therapy in Resectable GC/GEJC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-O17
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: GC/GEJC
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor; Docetaxel; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Intervention Model Description: Interventional Study Model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Mecapegfilgrastim plus Adebrelimab and FLOT (Experimental): Mecapegfilgrastim：（6 mg, HD, d3） Adebrelimab （1200 mg，iv d1） Docetaxel（50 mg/m2 iv gtt d1） Oxaliplatin （85 mg/m2 iv gtt d1） 5- fluorouracil, leucovorin （200 mg/m2 iv gtt d1） for 4 cycles (every 2 weeks) before surgery.
  Interventions: Drug: Mecapegfilgrastim; Drug: Adebrelimab; Drug: Docetaxel; Drug: Oxaliplatin; Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin (LV)
- Arm B: Adebrelimab plus FLOT (Experimental): Adebrelimab （1200 mg，iv d1） Docetaxel（50 mg/m2 iv gtt d1） Oxaliplatin （85 mg/m2 iv gtt d1） 5- fluorouracil, leucovorin （200 mg/m2 iv gtt d1） for 4 cycles (every 2 weeks) before surgery.
  Interventions: Drug: Adebrelimab; Drug: Docetaxel; Drug: Oxaliplatin; Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin (LV)

INTERVENTIONS:
Drug: Mecapegfilgrastim — 6 mg,HD d3,every 2weeks (Q2W)
  Arms: Arm A: Mecapegfilgrastim plus Adebrelimab and FLOT
Drug: Adebrelimab — Adebrelimab：1200 mg，iv d1，every2 weeks (Q2W)
Drug: Docetaxel — Docetaxel：50 mg/m2 iv gtt d1，every 2 weeks (Q2W)
Drug: Oxaliplatin — Oxaliplatin ：85 mg/m2 iv gtt d1，every2 weeks (Q2W)
Drug: 5-Fluorouracil (5-FU) — 5-FU ：2600 mg/m2 ，intravenous infusion， 24h ，d1，every 2 weeks (Q2W)
Drug: Leucovorin (LV) — LV：200 mg/m2 iv gtt d1，every 2 weeks (Q2W)

SUMMARY:
This study is a prospective, randomized ，multicencter, phase II clinical trial that aims to enroll patients with locally advanced gastric adenocarcinoma who have not received any prior treatment and are candidates for surgery. The purpose of this study is to assess the safety and efficacy of Mecapegfilgrastim Combined With Adebrelimab and 5- fluorouracil, leucovorin, oxaliplatin and docetaxel (FLOT)） as Neoadjuvant Therapy in Resectable gastric and gastroesophageal junction cancer

DETAILED DESCRIPTION:
After being informed about the study and potential risks, patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomly divided into trial group A and trial group B: Trial group A receive the combination therapy of Mecapegfilgrastim combined with Adebrelimab and FLOT, and trial group B receive the combination therapy of Adebrelimab combined with FLOT, two weeks a cycle, surgery was performed after 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects aged 18-75 years (including 18 and 75 years old);
* 2.Subjects who understand the study procedures and content, and voluntarily sign the written informed consent form;
* 3.Subjects with HER2-negative or HER2 status unknown gastric or gastroesophageal junction adenocarcinoma, clinically staged as T3-4a/N+M0 locally advanced gastric cancer by ultrasound gastroscopy, CT/MRI and other imaging evaluations.
* 4.Subjects who have not received prior systemic therapy.
* 5.Subjects with Eastern Cooperative Oncology Group Performance Status score (ECOG PS score): 0-1;
* 6.Subjects with life expectancy ≥ 12 months;
* 7.Subjects with good major organ function, that is, the relevant investigation indicators within 14 days before enrollment meet the following requirements: haemoglobin ≥ 90 g/L ; neutrophil count > 1.5 × 109/L; platelet count ≥ 100 × 109/L; total bilirubin ≤ 1.5 × ULN (upper limit of normal); alanine transaminase (ALT) or aspartate transaminases (AST) ≤ 2.5 × ULN; endogenous creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula); cardiac ultrasound doppler assessment: left ventricular ejection fraction (LVEF) ≥ 50%;
* 8.Subjects with thyroid function indicators: thyroid stimulating hormone (TSH), free thyroxine (FT3/FT4) within the normal range or with slight and clinically insignificant abnormalities;
* 9.Subjects weighing more than 40 kg, or with BMI > 18.5;

Exclusion Criteria:

* 1.Subjects with a history of or concurrent with other tumors malignant, except for cured early-stage tumors, including basal cell carcinoma of the skin and carcinoma in situ of the cervix, and early-stage tumors such as stage I lung cancer and stage I rectal cancer that have received radical treatment and are judged by the investigator not to affect the subject's life in the short term.
* 2.Subjects who have participated in other drug clinical studies within 4 weeks;
* 3.Subjects with a history of haemorrhage, the severity of any grade ≥ 3 haemorrhage event according to CTCAE 5.0 criteria within 4 weeks prior to screening;
* 4.Prior to screening, there were known highly suspected distant metastases, such as suspected peritoneal nodules, suspected cancerous ascites, and no laparoscopic confirmation;
* 5.Subjects with hypertension that cannot be well controlled with single-drug therapy (blood pressure systolic > 140 mmHg, blood pressure diastolic > 90 mmHg); subjects with a history of unstable angina pectoris; subjects newly diagnosed with angina pectoris within 3 months before screening or with myocardial infarction within 6 months before screening; arrhythmia (including QTcF: male ≥ 450 ms, female ≥ 470 ms) requiring long-term use of antiarrhythmic drugs and New York Heart Association class ≥ II cardiac insufficiency;
* 6.Subjects with long-term unhealed wounds or incompletely healed fractures;
* 7.Subjects whose imaging shows that the tumor has invaded the periphery of major blood vessels, or the investigator judges that the subject's tumor has a very high possibility of invading major blood vessels during treatment, causing fatal haemorrhage;
* 8.Subjects with abnormal coagulation function and haemorrhagic diathesis (must meet the following criteria within 14 days before enrollment: INR within the normal range without the use of anticoagulants); subjects treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues; low-dose warfarin (1 mg orally, once daily) or low-dose aspirin (daily dose not exceeding 100 mg) is allowed for prophylactic purposes, provided that the international normalized ratio (INR) of prothrombin time is ≤ 1.5;
* 9.Subjects with a history of arterial/venous thrombotic events within 6 months prior to screening, such as cerebrovascular accident (including transient ischaemic attack), deep vein thrombosis (excluding venous thrombosis caused by previous chemotherapy catheterization that has been judged to be cured by the investigator) and pulmonary embolism, etc.;
* 10.Subjects whose urinalysis test showing protein urine ≥ ++ and confirmed 24-hour protein urine quantification > 1.0 g;
* 11.Subjects with a history of immune targeted therapy;
* 12.Subjects with a history of immunodeficiency, or suffering from other acquired or immunodeficiency congenital diseases, or history of organ transplant;
* 13.Subjects with pneumonia, non-infectious pneumonia, interstitial pneumonia and other subjects who need to use corticosteroids;
* 14.Subjects with a history of severe chronic autoimmune diseases, such as systemic lupus erythematosus; a history of inflammatory bowel disease such as ulcerative enteritis, Crohn's disease; a history of chronic diarrheal diseases such as irritable bowel syndrome; a history of nodular disease or tuberculosis; active hepatitis B, hepatitis C, and HIV infection; well-controlled non-serious immune diseases such as dermatitis, arthritis, and psoriasis can be enrolled. Subjects with a hepatitis B virus titer < 2000 copy/mL can be enrolled.
* 15.Subjects with hypersensitivity to humanized or murine monoclonal antibodies;
* 16.Subjects with a history of mental drug abuse who are unable to abstain or who have a mental disorder;
* 17.Subjects who do not follow doctor's advice, do not take medicine as prescribed, or have incomplete data, which may affect the judgment of efficacy or safety;
* 18.Subjects with serious concomitant diseases that, in the judgment of the investigator, endanger the subject's safety or affect the subject's completion of the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | From enrollment to the end of treatment at 12 weeks
  The pCR refers to the proportion of subjects with no residual tumor cells in the primary lesion based on Becker Grade 1a.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | From enrollment to the end of treatment at 12weeks
  The proportion of subjects with resectable gastric cancer after neoadjuvant therapy who have less than 10% residual tumor cells in the primary lesion.
R0 Resection Rate | From enrollment to the end of treatment at about 12 weeks
  The R0 resection rate refers to the proportion of subjects with resectable gastric cancer who complete R0 resection in the total number of subjects operated. R0 resection refers to microscopically negative margins.
Event-free Survival (EFS) | 24 months
  The EFS refers to the time from the date of the random enrollment to disease progression, recurrence, or death (whichever occurs first).
Overall Survival (OS) | 36 months
  The OS refers to the time from the date of the random enrollment to death from any cause. For subjects who are still alive at the time of the last follow-up, OS is censored at the time of the last follow-up. For subjects lost to follow-up, their OS is censored at the last confirmed alive time before loss to follow-up. The censored OS is defined as the time from the date of the first dose to the time of censoring.
Chemotherapy completion rate | 8 weeks
  The proportion of patients who completed 4 cycles of FLOT chemotherapy in the total number of enrolled patients

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No